CLINICAL TRIAL: NCT05691543
Title: A Modified Technique in Sacrospinous Fixation Using Posterior Vaginal Wall Flap for Treatment of Apical Genital Prolapse
Brief Title: Modified Technique in Sacrospinous Fixation for Treatment of Apical Genital Prolapse
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: SSF
Record Dates: First submitted 2022-12-14; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Genital Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients with symptomatic Stage II , III and Stage IV Apical Prolapse (diagnosed by pop Q test)
  Interventions: Procedure: sacrospinous fixation Using Posterior Vaginal wall flap

INTERVENTIONS:
Procedure: sacrospinous fixation Using Posterior Vaginal wall flap — * Identification of the sacro spinous ligament.
  * Insertion of the sacrospinous stitch. Using a long - handled needle holder, a J - shaped Ethibond suture is placed 2 - 3 cm medial to the right ischial spine. Using posterior vaginal wall flap (rectangular flap )will be incised and retracted Superior to the right , the stitch of sacro spinous ligament will be attached to the flap not the vault after adjusting its size , then the sit . The stitch should be placed through and not around the ligament. The application of firm traction to the suture length will test the correctness of its placement. A second suture is inserted for additional support. We may do it directly or by using an alternative surgical instruments for placement of the suture include the knee scorpion. Per rectum examination should be undertaken to check for misplaced sutures.
  * Attachment of the sutures to the vaginal flap . The two sutures are then secured to the upper posterior aspect of the vaginal flap ,

SUMMARY:
Pelvic organ prolapse is one of the most common benign gynecological disorders and affects approximately 40% of women over 50 years of age. The causes of utero vaginal prolapse are pregnancy, labor, obesity, increased intra-abdominal pressure, and weak pelvic floor structures

ELIGIBILITY:
Inclusion Criteria:

1- Symptomatic Stage II , III and Stage IV Apical Prolapse (diagnosed by pop Q test ) .

Exclusion Criteria:

1. Patients with medical disorders that may interfere with surgical interventions ( Like severe chest and heart diseases , renal and liver cell failure , bleeding tendency ) .
2. Patients with urinary incontinence ( excluded by history , examination & Urodynamics)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with symptomatic Stage II , III and Stage IV Apical Prolapse (diagnosed by pop Q test)
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The difference of quality life score | 6 months
  this will be assessed before and after the surgery using

IPD SHARING:
Plan to Share IPD: No